CLINICAL TRIAL: NCT02228577
Title: A Study Assessing the Safety and Performance of the Transcend CyPass System Applier Model 241 for Implantation of the CyPass Micro-Stent in Subjects With Open Angle Glaucoma Who Underwent Cataract Surgery
Brief Title: Safety and Performance Study of the CyPass System Applier Model 241
Acronym: RePASS
Status: Completed | Type: Observational
Sponsor: Transcend Medical, Inc. (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Other Study IDs: TMI-14-01
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2016-10

CONDITIONS: Open Angle Glaucoma (OAG)
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective chart review of cases in which the CyPass Micro-Stent was implanted using the Model 241 Applier. The objective of this study is to characterize and evaluate the safety of the Model 241 Applier when used for CyPass Micro-Stent implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of OAG
2. CyPass Micro-Stent implantation (using the CyPass system 241) following uncomplicated phacoemulsification cataract removal and intraocular lens implantation

Exclusion Criteria:

1. Diagnosis of acute angle closure, traumatic, congenital, malignant, uveitic or neovascular glaucoma
2. Prior incisional glaucoma surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with OAG who underwent combination cataract/glaucoma surgery and received the CyPass Micro-Stent using the CyPass Applier Model 241
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Ocular adverse events in the study eye | Intraoperatively though the first 3 postoperative months

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik for Augenheilkunde - Dietrich Bonhoeffer Klinikum, Neubrandenburg, Germany

IPD SHARING:
Plan to Share IPD: No